CLINICAL TRIAL: NCT00801567
Title: A Magnetic Resonance Spectroscopy Study of Change in Brain Bioenergetics in Bipolar Disorder in Response to Photic Stimulation
Brief Title: Change in Brain Bioenergetics in Bipolar Disorder in Response to Photic Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of essential Co-Investigator from McLean Hospital
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director of Translational Neuroscience Research, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008-P-001958
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder; Schizophrenia; Healthy Controls
Keywords: Bipolar disorder; Schizophrenia; Healthy volunteer; Brain imaging; Photic stimulation
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects will receive the intervention (MRS scan).
  Interventions: Device: Magnetic resonance spectroscopy (MRS)

INTERVENTIONS:
Device: Magnetic resonance spectroscopy (MRS) — 90-minute magnetic resonance scan.

SUMMARY:
This study aims to gather additional information to support the theory that bipolar disorder is due to cellular (mitochondrial) dysfunction. To test this theory adults with bipolar disorder who are not currently symptomatic will receive a one-time brain scan (magnetic resonance spectroscopy [MRS] scan) with light stimulation. To test whether any MRS findings are specific to bipolar disorder, healthy controls and adults with schizophrenia will also be included in this study.

DETAILED DESCRIPTION:
This study will include males and females between the ages of 18 and 55 years. Participants will include adults with stable bipolar disorder or schizophrenia as well as healthy controls. The study involves a one-time visit that includes a clinical evaluation, laboratory tests, and a magnetic resonance scan that will last approximately 90 minutes. The procedures can also be separated into two study visits, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Male of female
* 18-55 years
* Bipolar, currently euthymic OR schizophrenia, stable, OR healthy control with no history of psychiatric illness
* On stable medication with no changes in the two weeks prior to enrollment

Exclusion Criteria:

* History of substance abuse or dependence within 3 months of enrollment
* Positive urine drug screen
* Significant medical or neurological illness
* Pregnancy
* Any contraindication to magnetic resonance scanning, including claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in brain levels of phosphocreatine (PCr), beta-nucleoside triphosphate (B-NTP), and intracellular pH (pHi). | 42 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States